CLINICAL TRIAL: NCT01095211
Title: Effect of B-Vitamins on Cognitive Function in Elderly People
Brief Title: B-vitamins Treatment for Improvement of Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Collaborators: Geriatrische Rehaklinik (Unknown)
Responsible Party: Dr. Eckert, Kreiskrankenhaus St. Ingbert GmbH
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Elderly St.Ingbert
Record Dates: First submitted 2010-03-29; First posted 2010-03-30 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Cognitive Function; Metabolic Improvements
Keywords: folic acid; homocysteine; MMSE scores; methyl malonic acid; betaine
MeSH Terms: interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- B-Vitamins (Active Comparator): folic acid, cobalamin, vitamin B6
  Interventions: Drug: B-vitamin complex
- placebo (Placebo Comparator): none of the vitamins (99.5% mannitol)
  Interventions: Drug: B-vitamin complex

INTERVENTIONS:
Drug: B-vitamin complex — 5 mg Folic acid, plus 1 mg cyanocobalamin and 40 mg vitamin B6) oral/ day. The placebo capsule contained 400 mg of mannitol: aerosil (99.5: 0.5). In addition, 1 mg/s.c cyanocobalamin daily
  Other Names: no other names

SUMMARY:
Observation studies documented a correlation between plasma concentrations of homocysteine and cognitive decline with age. The study hypothesis was that high doses of B-vitamins (as effective homocysteine lowering treatment) can improve cognitive function in elderly people.

DETAILED DESCRIPTION:
We performed a treatment with therapeutic doses of B-vitamins (folic acid, cobalamin, vitamin B6) for 45 days. We collected blood and tested the concentrations of the metabolic markers in blood at start, 3 weeks later and at the end. Cognitive function was tested at start and at the end.

ELIGIBILITY:
Inclusion Criteria:

* age > 65 years and glomerular filtration rate (GFR) > 35 ml/min

Exclusion Criteria:

* acute cancer or those who had coronary or cerebral event or thrombosis in the last 3 months were not eligible for the study.
* furthermore, people who had dementia (mini-mental state-examination scores MMSE < 15)
* those treated with B-vitamins
* those with renal insufficiency
* those receiving drugs that affect Hcy-metabolism (methotrexate, anti-epileptics, L-dopa) were not allowed to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 79 (Actual)
Dates: Start 2003-01; Primary Completion 2005-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Cognitive function | baseline and 45 days later

CONTACTS AND LOCATIONS:
Overall Officials: Rima Obeid, Principal Investigator — Department of Clinical Chemistry, University of Saarland
Locations (1):
- Dr. Eckert-, Sankt Ingbert, Saarland, Germany